CLINICAL TRIAL: NCT07250321
Title: Efficacy of Cerebellar Transcranial Direct Current Stimulation in Degenerative Ataxia. A Sham-controlled Clinical and Quantitative Analysis.
Brief Title: Efficacy of tDCS in Degenerative Ataxia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Massimiliano Pau, Full Professor of Bioengineering, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4642022/CE Study Code tDCS-ATX
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ataxia, Cerebellar; Ataxia - Genetic Diagnosis - Unknown; Ataxia, Spinocerebellar; Ataxias, Hereditary
Keywords: ataxia; tDCS; non-invasive brain stimulation; gait; upper limb; quantitative analysis
MeSH Terms: conditions — Cerebellar Ataxia; Spinocerebellar Ataxias; Spinocerebellar Degenerations; Ataxia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Sham-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): For sham stimulation the tDCS device delivered just a short ramp of current to let patients feel a skin sensation similar to those perceived by those actually treated.
  Interventions: Device: Sham (No Treatment)
- Real (Active Comparator)
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Anodal stimulation is delivered by a battery-driven stimulator (NeuroConn GmbH, 98693 Ilmenau, Germany) through a pair of saline-soaked surface sponge electrodes (7 x 5 cm2) producing a constant current of 2 mA for 20 min. An electroconductive gel is applied to the electrodes to reduce contact impedance and the electrodes are held in place using elastic gauzes Stimulation is preceded by a ramping up and ramping down for 20 sec at the beginning and at the end of each session, respectively. The anode is placed 2 cm under the inion and the cathode was placed over the right deltoid muscle. For sham stimulation the machine did not deliver any current after the ramping up, so both groups of patients could feel the same skin sensation.
  Other Names: Real
  Arms: Real
Device: Sham (No Treatment) — In the "Sham" arm, no current was delivered to the brain except for the initial few seconds
  Other Names: Sham
  Arms: Sham

SUMMARY:
Degenerative cerebellar ataxias are a group of rare diseases that cause gradual damage to the cerebellum, the part of the brain that controls balance and coordination. People with these conditions may have difficulty walking, keeping their balance, or coordinating movements. They may also experience vision problems, muscle stiffness, tremors, or changes in behavior, depending on the specific cause of the disease.

These disorders can greatly affect independence and quality of life, and unfortunately, there are currently no treatments that can stop or reverse the disease. Most care focuses on managing symptoms with physical therapy and medication.

Recently, a non-invasive brain stimulation technique called transcranial direct current stimulation (tDCS) has been studied as a possible way to improve movement and thinking in people with ataxia. However, results so far have been mixed, possibly because of differences in disease type, treatment methods, and how improvements are measured.

New technologies, such as motion sensors and movement analysis, are helping researchers better measure the effects of treatments on walking, balance, and hand movements in daily life.

The goal of the current study is to test whether stimulating the cerebellum with anodal tDCS can improve movement in people with different types of degenerative ataxia. The study will use both standard clinical scales and precise movement analysis to measure changes. In addition, researchers will use brain recordings (EEG) taken before and after stimulation to better understand how tDCS may work in the brain

DETAILED DESCRIPTION:
Degenerative cerebellar ataxias are a heterogeneous group of inherited and acquired disorders characterized by cerebellar atrophy and degeneration which leads to a wide range of clinical symptoms. Indeed, beside cerebellar symptoms such as gait ataxia, postural unbalance, dysmetria and nystagmus, patients may exhibit peripheral neuropathy, pyramidal and extrapyramidal signs and behavioural symptoms, depending on the aetiology of the disorder.

These disorders substantially affect autonomy and quality of life, yet effective disease-modifying or symptomatic treatments remain limited; their current management is largely supportive, including physical therapy and symptomatic pharmacological interventions.

Among non-pharmacological treatments, cerebellar transcranial direct current stimulation (tDCS), a non-invasive brain stimulation (NIBS) technique, has been employed in several studies with the aim to improve both motor and cognitive symptoms in different forms of ataxia, with conflicting results, so that, at present, it is not possible to determine its therapeutic potential with certainty. In this regard, it has been hypothesized that the large variability of clinical outcomes associated with such approach is due to several factors including, among the most relevant, the heterogeneity of ataxia aetiology, the significant differences in terms of protocols of stimulation and the lack of sensitive objective measures to be integrated with the scales traditionally employed in the clinical routine. Indeed, in the last years, quantitative analysis of movement (performed using either motion capture system or wearable inertial sensors) has shown to be a reliable approach to assess, in combination with clinical data, the existence and magnitude of possible positive effects induced by NIBS on basic motor functions (i.e., gait and balance) as well as to monitor real-world mobility and characterize physical activity patterns of people with ataxia.

The ability of cerebellar tDCS to influence the cerebellar-thalamus-cortical pathway has been demonstrated by the cerebellar-brain inhibition (CBI) TMS paradigm. Moreover, the cerebellar-cortical connectivity has been explored with NIBS combined with functional magnetic resonance imaging (fMRI) and EEG with online and offline paradigms. Several studies show that cerebellar NIBS is able to influence cortical oscillations and that an increase of beta power in frontal and parietal region is involved sensory-motor integration and motor control through the modulation of the cerebellar-thalums cortical circuit; the role of cortical gamma oscillation on motor activity following cerebellar stimulation is less characterized, but some evidence indicates that cortical gamma activity reflects excitatory action of the cerebellum on the motor thalamus and the motor cortex. However, in this case the results are controversial probably due to the heterogeneous methodological approaches.

Based on these observations, the aim of the present study was to assess the efficacy of cerebellar anodal tDCS in improving ataxia in different forms of degenerative ataxia with a sham-controlled approach, using validated clinical rating scales as well as quantitative techniques for human movement analysis focused on gait and upper limb functionality (i.e., hand-to-mouth task) as data on these motor tasks are already available for people with ataxia.

Moreover, in order to explore the mechanism underlying the therapeutic effect of cerebellar tDCS data obtained from resting state EEG before and after stimulation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* clinical, radiological and/or genetic diagnosis of cerebellar ataxia

Exclusion Criteria:

* presence of electrical stimulators (i.e., pacemaker), pregnancy, visual disfunction, cognitive decline, mild to moderate ataxic symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Modified International Cooperative Ataxia Rating Scale (MICARS) | Before the first tDCS session (T0) and after 10 sessions (2 weeks)
  The Modified International Cooperative Ataxia Rating Scale (MICARS) is a clinical tool used to assess and quantify the severity of ataxia, a neurological condition characterized by impaired coordination and balance. It is a streamlined version of the original International Cooperative Ataxia Rating Scale (ICARS), designed to improve ease of use, reliability, and sensitivity to clinical changes. MICARS evaluates key domains such as gait and posture, limb coordination, speech, and eye movements, providing a numerical score that reflects overall ataxia severity. It is commonly used in both clinical practice and research to monitor disease progression and treatment effects in patients with cerebellar ataxia and related disorders.

SECONDARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | Before the first tDCS session (T0) and after 2 weeks (10 sessions)
  The Scale for the Assessment and Rating of Ataxia (SARA) is a standardized clinical tool used to evaluate the severity and progression of ataxia. It consists of eight performance-based items that assess functions such as gait, stance, sitting, speech, and limb coordination (including finger-chase, nose-finger test, fast alternating hand movements, and heel-shin slide). Each item is scored on a defined scale, and the total score ranges from 0 (no ataxia) to 40 (most severe ataxia). SARA is valued for its simplicity, reliability, and sensitivity to change, making it widely used in both clinical trials and routine neurological assessments of cerebellar disorders.
Robertson Dysarthria profile | Befofe the first tDCS session and after 2 weeks (10 sessions)
  The Robertson Dysarthria Profile is a comprehensive clinical assessment tool used to evaluate and document speech difficulties associated with dysarthria, a motor speech disorder caused by neurological impairment. It examines key aspects of speech production, including respiration, phonation, articulation, resonance, and prosody, as well as the patient's intelligibility and communication effectiveness. The profile helps clinicians identify the type and severity of dysarthria, monitor changes over time, and plan targeted therapy. It is particularly useful in both diagnostic assessment and treatment planning for individuals with acquired or developmental speech motor disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) that will be collected throughout the trial will include all de-identified data relevant to the study's primary and secondary outcomes as well as demographic and clinical characteristics
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From January 2026 to December 2026
Access Criteria: Researcher and clinicians involved in ataxia studies

REFERENCES:
- [Derived] Sanna A, Pau M, Porta M, Pilia G, Secci V, Cartella E, Demattia A, Paribello A, Cossu G, Milia A, Tacconi P. Efficacy of Cerebellar Transcranial Direct Current Stimulation in Degenerative Ataxia. A Sham-Controlled Clinical and Quantitative Analysis. Cerebellum. 2026 Jan 14;25(1):11. doi: 10.1007/s12311-025-01952-6. PMID 41533249